CLINICAL TRIAL: NCT04421170
Title: Efficacy of Cognitive Behavioral Therapy-based Smartphone App for Smoking Cessation in China: a Study Protocol of a Randomized Controlled Trial
Brief Title: Efficacy of Smartphone App for Smoking Cessation in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Yanhui Liao, Principal Investigator, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20200129-33
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Cigarette Smoking; Smartphone App-based Smoking Cessation
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants from the intervention group will receive CBT based smoking cessation. It provides both mandatory information of evidence-based and guideline-based smoking cessation interventions, and optional information about quitting benefits, tips for quitting et al. The app will be available for the participants in the intervention group until 26-week post-quit date follow-up. After this period, the app will automatically stop the data collection, but they can continue to use it if they want. As the participants progressed through the study, smoking cessation related information will be gradually reduced until 12 weeks after quit date, and follow-up messages will be sent at 16, 20 and 26 weeks after quit date. Participants from intervention group can also seek for help at any time by text or WeChat, or make a phone call.
  Interventions: Behavioral: smartphone app for smoking cessation
- Control group (No Intervention): Participants from the control group will only receive information of thanking them for being in the study and reminding them of the time until their free month at the end of follow up. In order to measure the outcomes between two groups, continuous smoking abstinence, point prevalence of abstinence, how many cigarettes per day during the last week if they are still smoking will be checked at week 1, 2, 3, 4, 8, 12, 16, 20 and 26 points after quit date by ePRO software. Biochemically verified continuously abstinence will also be checked if they have reported continuous smoking abstinence at week 26 points after quit date.

INTERVENTIONS:
Behavioral: smartphone app for smoking cessation — Paticipants will receive 12-week app-based smoking cessation intervention with follow-up to 26 weeks.
  Arms: Intervention Group

SUMMARY:
This study aims to evaluate the efficacy of cognitive behavioral therapy (CBT)-based cigarette smoking cessation smartphone app for treatment seeking smokers in China.

ELIGIBILITY:
Inclusion Criteria:

1. Cigarette smokers (smoked more than 100 cigarettes in their lifetime, and currently smoke five or more cigarettes a day)
2. 25 years of age or older
3. Being able to read and write in Chinese
4. Owning a smartphone
5. Have experience of using apps
6. Expressing an interest in quitting smoking within the next month
7. Willing to provide informed consent to participate in the study

Exclusion Criteria:

1. Nonsmokers
2. Only use electronic cigarettes
3. Smokers without attempts to quit smoking
4. Participants with severe mental illness
5. Participants who had already started their quit attempt or using any smoking cessation treatment at the time of registration
6. Unable to use smartphone and apps
7. Unable to read and write in Chinese

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1289 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Biologically verified continuously smoking abstinence at week 26 | 26 weeks
  Participants in this study will be considered to be biologically verified continuously smoking abstinence if they report smoking no more than 5 cigarettes since the quit date and have an expired carbon monoxide concentration of less than 10 ppm (for local participants who will be able to go to the PI affiliated hospital) or a urine cotinine cutoff point of 200 ng/ml (cotinine urine dipsticks will be mailed to each participant's address, and test will be confirmed by video call and by family members) at week 26 (6 months) after quit date. This abstinence has been applied by the Society for Research on Nicotine and Tobacco (SRNT) (Hughes, Keely et al. 2003) and the 'Russell Standard' (West, Hajek et al. 2005).

SECONDARY OUTCOMES:
7-day point prevalence smoking abstinence | 26 weeks
  7-day Point prevalence of smoking abstinence: not even a puff of smoke, for the last seven consecutive days, at 1, 2, 3, 4, 8, 12, 16, 20 and 26 weeks.
Self-reported continuous smoking abstinence | 26 weeks
  Self-reported continuous smoking abstinence: a self-report of smoking ≤ 5 cigarettes from the past 1, 2, 3, 4, 8, 12, 16, 20 and 26 weeks.
Reductions in number of cigarettes smoked per day | 26 weeks
  Reductions in number of cigarettes smoked per day: will be assessed by comparing the number of cigarettes smoked per day at baseline and at 26 weeks. Cigarettes smoked per day: number of cigarettes smoked per day within seven days or the approximate total number of smoked cigarettes within seven days if not smoked daily.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhui Liao, MD, Principal Investigator — Department of Psychiatry, Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University
Locations (1):
- Yanhui Liao, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 1 month after publication.
Access Criteria: Yanhui Liao will review requests and criteria for reviewing requests

REFERENCES:
- [Derived] Chen S, Tang J, Wu C, Zhang G, Zhang J, Liao Y. Preliminary Efficacy of a Cognitive Behavioral Therapy-Based Smartphone App for Smoking Cessation in China: Randomized Controlled Pilot Trial. JMIR Form Res. 2024 Mar 18;8:e48050. doi: 10.2196/48050. PMID 38498030
- [Derived] Liao Y, Tang J. Efficacy of cognitive behavioural therapy-based smartphone app for smoking cessation in China: a study protocol of a randomised controlled trial. BMJ Open. 2021 Jan 13;11(1):e041985. doi: 10.1136/bmjopen-2020-041985. PMID 33441359